CLINICAL TRIAL: NCT00952159
Title: Validation of a New Method to Detect CYP2D6 Poor Metabolizers by Monitoring Seric Concentrations of O-demethyl-tramadol and Tramadol to Make a Ratio in Comparison With Genotyping in Post-operative Patients Treated With Intravenous Tramadol
Brief Title: CYTRAM (Cytochrome P450, Tramadol)
Acronym: CYTRAM
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Patrick MICHEL (research and strategy manager), Caen University Hospital
Other Study IDs: 2009-A00380-57; 09-013
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-07

CONDITIONS: Post-operative Patients Treated by Tramadol
Keywords: tramadol; CYP2D6; O-demethyl-tramadol; poor metabolizer; genotyping; phenotyping
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We propose to phenotype CYP2D6 in post-operative patients treated by tramadol by monitoring seric concentrations of O-demethyl tramadol and tramadol to make a ratio in comparision with genotype, and to find a threeshold to determine poor metabolizers. As already described, genotyping CYP2D6 will use a rapid detection method of the alleles implicated in poor metabolizer status (CYP2D6*3, *4, *5 et *6) in a caucasian population
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Not Poor metabolizer
  Interventions: Biological: Monitoring seric concentrations of O-demethyl-tramadol and tramadol
- Poor metabolizer
  Interventions: Biological: Monitoring seric concentrations of O-demethyl-tramadol and tramadol

INTERVENTIONS:
Biological: Monitoring seric concentrations of O-demethyl-tramadol and tramadol — The first aim of this study is the validation of monitoring seric concentrations of O-demethyl-tramadol and tramadol to make the ratio in order to detect CYP2D6 poor metabolizers in therapeutic situation, comparing the result with genotyping. The finding of a poor metabolizer status in a patient will make the choice of analgesic drugs easier, avoiding tramadol and codeine. The final objective of this research is to be able to determine the CYP2D6 phenotype in a patient treated by tramadol without a good analgesia. By a single take of blood and a rapid response, this method should be liked to improve pain management. Furthermore, CYP2D6 phenotyping is interesting for the patient because many other drugs depend on this way of metabolism.

SUMMARY:
Many methods to detect CYP2D6 poor metabolizers have been validated. Some of them are based on phenotyping (metabolism of dextromethorphan or debrisoquine) and some others on genotyping. Up to now, CYP2D6 pharmacogenetics has been restricted to the field of research, in spite of poor metabolizer profile concerns 5 to 10 % of caucasian population. Nevertheless, the polymorphism of CYP2D6 is responsible for the metabolism of many drugs, particularly of two opioids involved in pain management: codeine and tramadol, their metabolites representing the most effective part of the drug effect. So prescribing codeine or tramadol in a patient poor metabolizer for the CYP2D6 is likely to be ineffective in pain management.

O-demethyl-tramadol, the metabolite of tramadol via CYP2D6, is important to consider because its analgesic effect is 2 to 4 times more potent than tramadol.

The investigators propose to phenotype CYP2D6 in post-operative patients treated by tramadol by monitoring seric concentrations of O-demethyl tramadol and tramadol to make a ratio in comparison with genotype, and to find a threshold to determine poor metabolizers. As already described, genotyping CYP2D6 will use a rapid detection method of the alleles implicated in poor metabolizer status (CYP2D6*3, *4, *5 et *6) in a Caucasian population. Sampling will be executed at two times (H24 and H48 after surgery) and only with blood (three EDTA tubes) during the post-operative monitoring of the patients. This study is likely to include 320 post-operative patients treated with intravenous tramadol during one year in three university hospitals centers (CHU of Caen, Creteil and Rouen).

The first aim of this study is the validation of monitoring seric concentrations of O-demethyl-tramadol and tramadol to make the ratio in order to detect CYP2D6 poor metabolizers in therapeutic situation, comparing the result with genotyping. The finding of a poor metabolizer status in a patient will make the choice of analgesic drugs easier, avoiding tramadol and codeine. The final objective of this research is to be able to determine the CYP2D6 phenotype in a patient treated by tramadol without a good analgesia. By a single take of blood and a rapid response, this method should be liked to improve pain management. Furthermore, CYP2D6 phenotyping is interesting for the patient because many other drugs depend on this way of metabolism.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years, post-operative patient treated with intravenous tramadol
* Caucasian origin
* take of blood at H24 and H48 in the post-operative monitoring

Exclusion Criteria:

* patient having already been included in the study
* patient taking opioid drugs before surgery
* patient taking one or more drugs inhibiting the CYP2D6 before or during surgery
* pregnancy or breast feeding patients having one or more contraindications for taking tramadol in post-operative analgesia
* hepatocellular incapacity (TP < 70%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-operative patients treated by tramadol
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To phenotype CYP2D6 in post-operative patients treated by tramadol by monitoring seric concentrations of O-demethyl tramadol and tramadol to make a ratio in comparison with genotype, and to find a threshold to determine poor metabolizers. | H24 and H48 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Blandine de la Gastine, MD, Principal Investigator — University Hospital, Caen
Locations (4):
- France (4):
  - Private Clinic Saint-Martin, Caen
  - Caen University Hospital, Caen
  - Créteil University Hospital, Créteil
  - Rouen University Hospital, Rouen